CLINICAL TRIAL: NCT06812000
Title: Investigation of Incidence Rate of Post-stroke Seizure and Post-stroke Epilepsy in Patients Under Treatment With Alteplase and Correlated Factors
Brief Title: Post-stroke Seizure and Epilepsy Following Thrombolytic Therapy
Status: Completed | Type: Observational
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Associate professor of neurology, Mazandaran University of Medical Sciences
Other Study IDs: 17989
Record Dates: First submitted 2025-01-17; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Post-stroke Seizure; Post-stroke Epilepsy; Thrombolytic (t-PA) Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ischemic stroke who received alteplase: Patients with ischemic stroke who received thrombolytic therapy with alteplase
- Patients with ischemic stroke who did not receive alteplase: Patients with ischemic stroke who did not receive thrombolytic therapy

SUMMARY:
This retrospective cohort study was conducted by reviewing the records of consecutive patients referred to Bu Ali Sina Hospital from 2016 to 2023, who were hospitalized with a diagnosis of ischemic stroke. The records of all patients treated with intravenous alteplase during the above period were extracted, and the relevant characteristics were recorded in a questionnaire. In each year, patients with ischemic stroke who were not treated with alteplase but were hospitalized at the Bu Ali Center were selected in a similar number to patients who received alteplase in the same year, and the relevant information was extracted from their records and recorded in a questionnaire. The incidence of post-stroke seizures and epilepsy was determined in both groups, and the factors associated with their incidence were studied and compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke
* Treatment with IV alteplase

Exclusion Criteria:

* History of epilepsy
* Taking antiseizure medications
* Unavailable patients
* Unreliability of recorded patients' files

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke who were admitted between 2016 and 2023 in Bu Ali Sina hospital
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of post-stroke seizure | within 7 days following ischemic stroke onset
  Incidence rate of post-stroke seizure in patients who received alteplase compared to patients who did not receive alteplase.
Incidence rate of post-stroke epilepsy | 1 to 7 years following ischemic stroke onset
  Incidence rate of post-stroke epilepsy in patients who received alteplase compared to patients who did not receive alteplase.

SECONDARY OUTCOMES:
Factors related to post-stroke seizure occurrence | within 7 days following ischemic stroke onset
  Demographic factors are registered in the questionnaire based on the patients' files. The severity of ischemic stroke is determined by the National Institutes of Health Stroke Scale (NIHSS). Brain CT findings including territory of infarct, cortical involvement and hemorrhagic transformation are investigated by reviewing the CT scans and recording the results in the questionnaire. Correlation of each mentioned factor with post-stroke seizure occurrence will be assessed using statistical methods.
Factors related to post-stroke epilepsy occurrence | 1 to 7 years following ischemic stroke onset
  Demographic factors are registered in the questionnaire based on the patients' files. The severity of ischemic stroke is determined by the National Institutes of Health Stroke Scale (NIHSS). Brain CT findings including territory of infarct, cortical involvement and hemorrhagic transformation are investigated by reviewing the CT scans and recording the results in the questionnaire. Correlation of each mentioned factor with post-stroke epilepsy occurrence will be assessed using statistical methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Mazandaran University of Medical Sciences, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: Undecided